CLINICAL TRIAL: NCT06764277
Title: Mechanisms and Phenotypes of Hypertension in Patients in Chronic Hemodialysis
Status: Completed | Type: Observational
Sponsor: Bernardo Rodríguez Iturbe (Other)
Responsible Party: Sponsor-Investigator, Bernardo Rodríguez Iturbe, Researcher, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Organization: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Other Study IDs: NMM-4512-23-24-1
Record Dates: First submitted 2024-12-19; First posted 2025-01-08 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Arterial Hypertension; Hemodialysis
Keywords: hemodialysis; hypertension; inflammation; renin angiotensin system; sympathetic nervous system; interdialysis; Interdialytic weight gain
MeSH Terms: conditions — Hypertension; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples: Serum levels of angiotensin II, norepinephrine, copeptin, Peripheral blood: Ratio of monocytes + neutrophils / lymphocytes (MNLR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: There will be no intervention. Group A will be patients with ABP (ambulatory blood pressure) <130/80 mmHg (controlled hypertension)
  Interventions: Other: There will be no intervention
- Group B: There will be no intervention. Group B will be patients with ABP 130-139/80-89 mmHg (insufficiently controled hypertension)
  Interventions: Other: There will be no intervention
- Group C: There will be no intervention. Group C will be patients with ABP ≥140/90 mmHg (uncontrolled hypertension)
  Interventions: Other: There will be no intervention

INTERVENTIONS:
Other: There will be no intervention — There will be no intervention. This is an observational studies and 3 groups will be organized depending on the level of ABP in the interdialytic period

SUMMARY:
The goal of this study is to evaluate interdialytic blood pressure changes of the patients in chronic hemodialysis.

The main question to be answered is: What is the relative importance of weight gain, the renin angiotensin system, the sympathetic nervous system and inflammatory immune reactivity in the interdialytic hypertension of patients in chronic hemodialysis, The participants will have hemodynamic evaluation (cardiac output and peripheral vascular resistance) at the end of dialysis, ambulatory monitoring of blood pressure in the interdialytic period. Serum samples will be collected at the end of dialysis and before the start of the next dialysis, 2-3 days later.

DETAILED DESCRIPTION:
This is a prospective observational study that will study stable patients in the chronic hemodialysis program of the Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán" (INCMNSZ) patients. There will be no modifications in the dialysis prescriptions or treatments and the patients with inclusion criteria will be studied after and before their usual hemodialysis sesion.

* Weight changes will be studied after dialysis and before the next dialysis session (2-3 days later)
* Serum samples will be obtained at the end of dialysis and before the next session (2-3 days later).
* ultrasound estimation of cardiac output and peripheral vascular rersistance will be done after dialysis
* Ambulatory blood pressure (ABP) monitoring will be done in the interdialytic period (24-40 hours) between the end of dialysis and the next dialysis session.
* If possible there will be a predialysis study of bioimpedance.
* Associations of interdialytic weight gain, serum angiotensin II, copeptin levels (surrogate of arginine vasopressin) and norepinephrine levels with ABP, systolic and diastolic blood pressure before and after dialysis will be explored.
* Phenotypes of blood pressure (sustained hypertension, nocturnal and diurnal hypertension, dippers, non-dippers, extreme dippers and reverse dippers) determined by ambulatory monitoring will be studied in relation of levels of angiotensin II, inflammatory markers, copeptin and norepinephrine levels.

All serum levels will be determined by commercial ELISA kits

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 3 months in the chronic hemodialysis program in the INCMNSZ and assumed to remained in the program for longer than 3 months
* Stable patients with no change in medication 1 month prior to the study
* Unchanged drug therapy and dialysis prescription for >1 month prior to the studies
* Informed consent to participate in the study

Exclusion Criteria:

* Patients unable to give informed consent or withdrawal of informed consent to the study
* Patients with active infection
* Patients with prosthesis or pacemakers
* Patients with immunosuppressive treatment of more than 10mg Prednisone daily
* Prior nephrectomy
* incomplete collection of data specified in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participantes will be patients in the chronic hemodialysis program of the INCMNSZ assigned to the groups depending on the ambulatory blood pressure (ABP) monitoring: Group A (TA < 130/80 mmHg), group B (TA 130-139/80-89 mmHg and group C (TA > 140mmHg)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo RODRIGUEZITURBE, MD, PhD, Principal Investigator — Department of Nephrology, Instituto Nacional de Ciencias Medicas y Nutrición "Salvador Zubirán"
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Iturbe B. Autoimmunity in the Pathogenesis of Hypertension. Hypertension. 2016 Mar;67(3):477-83. doi: 10.1161/HYPERTENSIONAHA.115.06418. Epub 2015 Dec 7. No abstract available. PMID 26644240
- [Background] Fay KS, Cohen DL. Resistant Hypertension in People With CKD: A Review. Am J Kidney Dis. 2021 Jan;77(1):110-121. doi: 10.1053/j.ajkd.2020.04.017. Epub 2020 Jul 23. PMID 32712185
- [Background] Abais-Battad JM, Rudemiller NP, Mattson DL. Hypertension and immunity: mechanisms of T cell activation and pathways of hypertension. Curr Opin Nephrol Hypertens. 2015 Sep;24(5):470-4. doi: 10.1097/MNH.0000000000000146. PMID 26125645
- [Background] Agarwal R, Weir MR. Dry-weight: a concept revisited in an effort to avoid medication-directed approaches for blood pressure control in hemodialysis patients. Clin J Am Soc Nephrol. 2010 Jul;5(7):1255-60. doi: 10.2215/CJN.01760210. Epub 2010 May 27. PMID 20507951
- [Background] Rodriguez-Iturbe B, Pons H, Johnson RJ. Role of the Immune System in Hypertension. Physiol Rev. 2017 Jul 1;97(3):1127-1164. doi: 10.1152/physrev.00031.2016. PMID 28566539
- [Background] Neumann J, Ligtenberg G, Klein II, Koomans HA, Blankestijn PJ. Sympathetic hyperactivity in chronic kidney disease: pathogenesis, clinical relevance, and treatment. Kidney Int. 2004 May;65(5):1568-76. doi: 10.1111/j.1523-1755.2004.00552.x. PMID 15086894
- [Background] Kim KE, Onesti G, Schwartz AB, Chinitz JL, Swartz C. Hemodynamics of hypertension in chronic end-stage renal disease. Circulation. 1972 Sep;46(3):456-64. doi: 10.1161/01.cir.46.3.456. No abstract available. PMID 4561117
- [Background] Buckalew VM Jr, Berg RL, Wang SR, Porush JG, Rauch S, Schulman G. Prevalence of hypertension in 1,795 subjects with chronic renal disease: the modification of diet in renal disease study baseline cohort. Modification of Diet in Renal Disease Study Group. Am J Kidney Dis. 1996 Dec;28(6):811-21. doi: 10.1016/s0272-6386(96)90380-7. PMID 8957032
- [Background] Saad E, Charra B, Raj DS. Hypertension control with daily dialysis. Semin Dial. 2004 Jul-Aug;17(4):295-8. doi: 10.1111/j.0894-0959.2004.17330.x. PMID 15250921

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (ABP < 130/80 mmHg): Constituted by15 patients in the chronic hemodialisis program with ABP < 130/80 mmHg, and we measured interdialytic weight gain, cardiac output, systemic vascular resistance, blood pressure changes, interdialytic ambulatory blood pressure monitoring (ABPM) . Serum levels of angiotensin II, norepinephrin, copeptin and the ratio of monocytes + neutrophils / linphocytes (MNLR)
- Group B (ABP 130-139/80-89 mmHg): This group was constituted by patients with ABP 130-139/80-89 mmHg. They were 7 patients in the chronic hemodialisis program, and we measured blood pressure changes, interdialysis ambulatory blood pressure monitoring (ABPM) and interdialisis weight gain. Serum levels of angiotensin II, norepinephrin, copeptin and the ratio of monocytes + neutrophils / lymphocytes (MNLR).
- Group C (ABP ≥ 140/90 mmHg): Constituted by 10 patients in the chronic hemodialisis program, with ABP ≥ 140/90 mmHg. We measured blood pressure changes, interdialysis ambulatory blood pressure monitoring (ABPM) and interdialisis weight gain. Serum levels of angiotensin II, norepinephrin, copeptin, and the ratio of monocytes + neutrophils / linphocytes (MNLR)
Period: Overall Study
Arm/Group | Group A (ABP < 130/80 mmHg) | Group B (ABP 130-139/80-89 mmHg) | Group C (ABP ≥ 140/90 mmHg)
Started | 15 (participants with ABP <130/80 mmHg) | 7 (participants) | 10 (participants)
Completed | 15 (participants) | 7 (participants) | 10 (participants)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Inclusion criteria: >18 years, >6 months in chronic hemodialysis, estable clinical conditions with no evidence of infection, or changes in medications, dialysis characteristics are not modified in the last months and sign informed consent to participate in the study.
  Exclusion criteria: previous nephrectomy, administration of eritropoyetin at the end of dialysis at the end of the stydu, participation of patient in other study, requiered a clinical intervention and incomplete collection of data
Groups:
- Group A (ABP < 130/80 mmHg): We observed 15 patients in the chronic hemodialysis program with ABP < 130/80 mmHg, and we measured blood pressure changes, interdialytic ambulatory blood pressure monitoring and interdialytic weight gain. Serum levels of angiotensin II, norepinephrine, copeptin, and the ratio of monocytes + neutrophils / lymphocytes (MNLR).
- Group B (ABP 130-139/80-89 mmHg): We observed 7 patients in the chronic hemodialysis program with ABP 130-139/80-89 mmHg , and we measured blood pressure changes, interdialytic ambulatory blood pressure monitoring and interdialysis weight gain. Serum levels of angiotensin II, norepinephrine, copeptin, and the ratio of monocytes + neutrophils / lymphocytes (MNLR).
- Group C (ABP ≥ 140/90 mmHg): We observed 10 patients in the chronic hemodialysis program with ABP ≥ 140/90 mmHg and we measured blood pressure changes, interdialytic ambulatory blood pressure monitoring and interdialytic weight gain. Serum levels of angiotensin II, norepinephrine, copeptin, and the ratio of monocytes + neutrophils / lymphocytes (MNLR).
- Total: Total of all reporting groups
Arm/Group | Group A (ABP < 130/80 mmHg) | Group B (ABP 130-139/80-89 mmHg) | Group C (ABP ≥ 140/90 mmHg) | Total
Number analyzed (Participants) | 15 | 7 | 10 | 32
Age, Continuous [Mean (Full Range); unit: years] | 38 [23 to 68] | 44 [33 to 72] | 35 [26 to 67] | 39 [23 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 5 | 19
  Male | 3 | 5 | 5 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — All parcipants were from Mexico City. Volunteers from the chronic hemodialysis program
  participants
    Mexico | 15 | 7 | 10 | 32
Cardiac output [Mean (Standard Deviation); unit: L/min] — Cardiac output (CO) =systolic volume x heart rate. Determined by 2 experienced observers using a Siemens Acuson P500 ultrasound equipment with a phased array transducer . Systolic volume was calculated with the velocity time integral of the flow of the left ventricle outflow tract of the aortic area.
  L/min | 3.88 (0.99) | 4.10 (0.77) | 4.55 (1.21) | 4.25 (0.34)
Hypertension Phenotypes [Count of Participants; unit: Participants] — Definitions:
  normal dippers when the blood pressure falls at night between 10-20% non- dippers when the blood pressure falls at night less than 10% reverse-dippers when the blood pressures increases during sleep instead of falling.
  extreme dippers when the blood pressure falls at night more than 20% Population: Number of participants indicate the participants analized in groups A, B and C (all members of each group (total of 32 participantes). The number of deepers, non-deepers, extreme deepers and reverse deepers was different in each group but the total number is also 32
  Participants
    Dippers | 5 | 3 | 1 | 9
    Non-dippers | 5 | 2 | 4 | 11
    Extreme Dippers | 1 | 0 | 0 | 1
    Reverse-dippers | 4 | 2 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Output
Description: Cardiac output (systolic volume x heart rate) was determined by 2 experienced observers using a Siemens Acuson P500 ultrasound equipment with a phased array transducer . Systolic volume was calculated with the velocity time integral of the flow of the left ventricle outflow tract of the aortic area.
Time Frame: Each participant was studied once 1-3 hours after dialysis ended
Population: Patients were mexicans of both sexes of mixed (undetermined) race and ethnicity
Measure: Mean (Standard Error); unit: L/min
Groups:
- Group A: Patients with ambulatory blood pressure (ABP) monitoring <130/80 mmHg
- Group B: Patients with ABP 130-139/80-89 mmHg
- Group C: Patients with ABP ≥140/90 mmHg
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 7 | 10
L/min | 3.9 (0.26) | 4.10 (0.29) | 4.6 (0.38)

2. Primary Outcome: Interdialytic Weight Change
Description: The weight was determined in 2 ocassions: first, immediately after dialysis and second, 2-3 days later, before the next dialysis. The weight change in this interval is expressed as percentage change of the second measure in relation to the first measure.
Time Frame: Interdialytic weight change was studied once, by the difference between the weight at the end of dialysis and the weight 2-3 days later, before the next dialysis.
Population: Patients were mexicans of both sexes and mixed (undetermined) race and ethnicity
Measure: Mean (Standard Error); unit: percentage change
Groups:
- Group A: Constituted by 15 patients with ABP < 130/80 mmHg
- Group B: constituted by 7 patients with ABP 130-139 mmHg
- Group C: Constituted by 10 patients in the chronic hemodialisis program with ABP ≥ 140/90 mmHg
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 7 | 10
percentage change | 2.90 (0.37) | 3.22 (0.63) | 2.98 (0.53)

3. Primary Outcome: Systemic Vascular Resistance
Description: Systemic vascular resistance was calculated using MediCalcR using the mean arterial pressure (MAP), the central venous pressure (CVP) anf the cardiac output (CO) and the equation: SVR=[(MAP-CVP)x79.92]/CO. Cardiac output (CO= systolic volume x heart rate) and central venous pressure were determined by 2 experienced observers using a Siemens Acuson P500 ultrasound equipment with a phased array transducer. Systolic volume was calculated with the velocity time integral of the flow of the left ventricle outflow tract of the aortic area.
Time Frame: Systemic vascular resistance was determined once in the participants 1-3 hours after dialysis
Population: All the participants were mexicans of both sexes and mixed (undetermined) race and ethnicity
Measure: Mean (Standard Error); unit: dynes*s/cm˄5
Groups:
- Group A: interdialytic ambulatory blood pressure <130/80 mmHg (6 normotensive patients and 9 patients with controlled hypertension)
- Group B: interdialytic ambulatoryblood pressure 130-139/80-89 mmHg (7 patients with insufficiently controlled hypertension
- Group C: Interdialytic ambulatory blood pressure ≥ 140/90 mmHg (10 patients with uncontrolled hypertension).
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 7 | 10
dynes*s/cm˄5 | 1513 (114.6) | 2045 (161.0) | 1751 (187)

4. Secondary Outcome: Angiotensin II Serum Levels
Description: Angiotensin serum levels (pg/ml) were determined once at the end of the interdialytic period, before dialysis, using ELISA (my BioSource Cat.# MBS703599)
Time Frame: Each participant was studied once. Serum samples taken before dialysis
Population: The participants were mexican of both sexes and mixed (undetermined) race and ethnicity
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- Group A: Constituted by 15 patients with ABP <130/80
- Group B: Constituted by 7 patients with ABP 130-139 mmHg .
- Group C: Constituted by 10 patients with ABP ≥140/90 mmHg
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 7 | 10
pg/ml | 105.3 (12.9) | 158.3 (43.8) | 231.5 (40.4)

5. Secondary Outcome: Monocyte+Neutrophiles/Lymphocyte Ratio (MNLR)
Description: Monocyte+Neutrophile/lymphocyte ratio obtained from peripheral blood counts in samples taken before dialysis (following the end of the interdialytic period).
Time Frame: Each participant was studied once. Blood samples taken before dialysis (following the end of the interdialytic period).
Population: Participants were mexicans of mixed (undetermined) race
Measure: Mean (Standard Error); unit: ratio
Groups:
- Group A: Constituted by 15 patients with ABP <130/80 mmHg
- Group B: Constituted by 7 patients with ABP 130-139/80-89 mmHg
- Group C: onstituted by 10 patients with ≥140/90 mmHg
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 7 | 10
ratio | 0.88 (0.13) | 0.73 (0.09) | 1.11 (0.13)

6. Secondary Outcome: Serum Norepinephrine Levels
Description: Interdialytic serum norepinephrine levels determined in blood samples obtained before dialysis (end of interdialytic period) using ELISA (ABCAM, Cat. # AB287789);
Time Frame: Each participant was studied once. Serum samples taken before dialysis
Population: The studies were done at the end of the interdialytic period. Samples taken before the next dialysis
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Group C: Constituted by 10 patients with ≥140/90 mmHg.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 15 | 7 | 10
pg/ml | 81.4 [68.5 to 87.4] | 82.4 [66.5 to 165.4] | 82.6 [74.9 to 259.0]

7. Secondary Outcome: Serum Copeptin Levels
Description: The copeptin levels (surrogate for arginine vasopressin) were measured before dialyisis (end of the interdialytic period) using ELISA (Bio-techne/NovusBiological, Cat, # NBP2-69822)
Time Frame: Each participant was studied once. Serum samples taken before dialysis
Population: Mexican mixed population of undetermined race
Measure: Mean (Standard Error); unit: pmol/L
Groups:
- Group B: Constituted by 7 patients who had ABP 130-139/80-89 mmHg.
- Group C: Constituted by 10 patient with ABP ≥140/90 mmHg.
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 11 | 6 | 9
pmol/L | 14.6 (1.09) | 10.3 (0.92) | 13.0 (1.56)

8. Secondary Outcome: Hypertension Phenotypes
Description: Interdialytic ambulatory blood pressure determined during 24-44 hours using Space Labs Health Care, model 90217A and Contec ABPM50 equipment. Determinations every 30 minutes during daytime and every hour during the night. We are here reporting the phenotypes in the total number of participants (n=32) instead that in each group (groups A n=15, B n=7 and C n=10) because our main interest was to determine the incidence of each phenotyte in stable patients treated with chronic dialysis, rather than in each group that, individually, had few patients
Time Frame: Each participant was studied once. Ambulatory blood pressure was monitored or 24-44 hours during the interdialytic perdiod starting 1-3 hours after dialysis
Population: The number of dippers, non-dippers, extreme dippers and reverse dippers were studied in all participants (n=32) .
Measure: Count of Participants; unit: Participants
Groups:
- Blood Pressure Dipper: Nocturnal reduction 0f blood presure of 10-20%
- Excesive Dipper: Nocturnal blood pressure reduction of >20 % of daytime pressure
- Non-dipper: Nocturnal blood pressure reduction <10% of day time blood pressure
- Reverse Dipper: Nocturnal blood pressure higher than diurnal blood pressure
Arm/Group | Blood Pressure Dipper | Excesive Dipper | Non-dipper | Reverse Dipper
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants | 8 | 1 | 13 | 10

ADVERSE EVENTS:
Time Frame: The observational study was performed through 1 to 3 days and no adverse events were reported.
Description: The observational study was performedThe observational study was performed through 1 to 3 days and no adverse events were reported or death.
Groups:
- Group 1 (TA < 130mmHg): We observed 15 patients in the chronic hemodialysis program, and we measured blood pressure changes, interdialytic ambulatory blood pressure monitoring (ABPM) and interdialytic weight gain. Serum levels of angiotensin II, norepinephrine, copeptin, tumor necrosis factor alpha (TNF-a), and the ratio of monocytes + neutrophils / lymphocytes.
- Group 2 (TA 130-139mmHg): We observed 7 patients in the chronic hemodialysis program, and we measured blood pressure changes, interdialytic ambulatory blood pressure monitoring (ABPM) and interdialyticweight gain. Serum levels of angiotensin II, norepinephrine, copeptin, TNF-a, and the ratio of monocytes + neutrophils / lymphocytes.
- Group 3 (TA > 140): We observed 10 patients in the chronic hemodialysis program, and we measured blood pressure changes, interdialytic ambulatory blood pressure monitoring (ABPM) and interdialytic weight gain. Serum levels of angiotensin II, norepinephrine, copeptin, TNF-a, and the ratio of monocytes + neutrophils / lymphocytes.
Arm/Group | Group 1 (TA < 130mmHg) | Group 2 (TA 130-139mmHg) | Group 3 (TA > 140)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 0/15 | 0/7 | 0/10

LIMITATIONS AND CAVEATS:
1) Potential effects of antihypertension drug therapy (observational study) may not be completely discarded. 2)Only 32 patients in only one recruitment center. Further studies are required to validate the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT06764277/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT06764277/SAP_001.pdf
  • Informed Consent Form (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT06764277/ICF_002.pdf